CLINICAL TRIAL: NCT02840981
Title: Obese Patients Adhering to Mediterranean Diet Show Less Reduced Circulating Levels of Sirtuin 4
Brief Title: Adherence to the Mediterranean Diet and Circulating Levels of Sirtuin 4 in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Prof. Silvia Savastano, Researcher/Adjunct Professor, Federico II University
Other Study IDs: 5/14
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Mediterranean Diet; Nutrition; Sirtuin 4; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The Mediterranean diet (MD), a healthy dietary pattern based on some common dietary characteristics in Mediterranean countries, is associated with high antioxidant capacity linked to the low saturated fat intake that might contribute to reduce free fatty acid (FFA) availability and oxidation in mitochondria, thus reducing the production of the reactive oxygen species (ROS) superoxide, and promoting cellular health. To assess the adherence to the MD, a simple 14-item questionnaire had been tested in different settings by the PREDIMED (PREvención con DIeta MEDiterránea) multicenter, randomized, primary prevention trial. On the other hand, to allow a more an accurate measurement of the actual macro and micronutrient intakes, including dietary anti-oxidant micronutrients, the 7-day food records is considered as the "gold standard" of self-administered food frequency questionnaires.

Circulating levels of Sirtuin 4 (Sirt4), part of a complex of proteins that control diverse biological processes, including lipid metabolism, are low in obese patients, as a possible attempt to decrease fat oxidative capacity and mitochondrial ROS production, however promoting ectopic liver fat storage.

The phase angle (PA), a measure determined by bioelectrical impedance analysis (BIA), and the visceral adiposity index (VAI), a gender-specific mathematical index based on simple anthropometric and metabolic parameters, represent well-validated, reliable and widely used markers of cellular health and ectopic adipose distribution and function, respectively. The fatty liver index (FLI) is a surrogate measure for fatty liver recently proposed as an independent predictor for diabetes mellitus.

Aim of the present study was to investigate in adult obese individuals the levels of Sirt4 according to the adherence to the MD evaluated by PREDIMED questionnaire, focusing on the possible association with single dietary components evaluated by 7-day food records, and to evaluate the association between circulating levels of Sirt4 and PA, as marker of cellular health, VAI, as index of adipocyte dysfunction, and FLI, as a predictor of fatty liver.

ELIGIBILITY:
Inclusion Criteria:

* Adult obese subjects

Exclusion Criteria:

* Hypocaloric diet in the last three months or specific nutritional regimens, including vegan or vegetarian diets;
* Presence of liver or renal failure, cancer, and acute or chronic inflammatory diseases based on a complete medical examination and laboratory investigations (psoriasis, rheumatoid arthritis and chronic obstructive pulmonary disease);
* Occasional or current of use of drugs affecting β-oxidation, including non-steroidal anti-inflammatory drugs, α-lipoic acid, valproic acid
* Use of weight loss medication or lipid-lowering drugs
* Altered thyroid hormone function tests or thyroid hormone treatment or altered somatotropic axis
* Alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders (DSM)-V diagnostic criteria
* Vitamin/mineral or antioxidant supplementation
* Subjects dropped out from the study since they refused to undergo full laboratory-instrumental examinations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 257 consecutive obese subjects visiting the out-patient Obesity Unit of the Section of Endocrinology, University of Naples Federico II
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Adherence to Mediterranean Diet by Predimed Questionnaire | December 2013 to September 2015
Circulating Levels of Sirtuin 4 by ELISA method | December 2013 to September 2015
Obesity by Body Mass Index | December 2013 to September 2015